CLINICAL TRIAL: NCT00449826
Title: Risk Stratification of Non ST Elevation ACS With Computed Tomographic Angiography (REACT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Benjamin Chow, Dr Benjamin Chow, Ottawa Heart Institute Research Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UOHI 2006361-01H
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Acute Coronary Syndrome; Non-ST-Elevation Myocardial Infarction; Unstable Angina
Keywords: ACS; Unstable Angina; NSTEMI
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: Computed Tomographic Angiography — CT scan

SUMMARY:
The purpose of this project is to examine the effectiveness of computed tomographic angiography (CTA) in patients with non-ST elevation acute coronary syndrome (NSTE-ACS). People who are hospitalized with this situation often require an angiogram to assess the heart and its arteries.

Recent advancements in technology have enabled CTA to clearly define coronary artery anatomy with great accuracy and to guide treatment strategies in select patient populations. We are investigating that CTA may be used, as an alternative to conventional angiograms, for the risk stratification of patients with high risk NSTE-ACS.

Patients eligible for the study will be high risk NSTE-ACS and awaiting an angiogram. Enrolled patients will undergo CTA prior to the angiogram. With each CTA the patient will be injected with a small dose of an X-ray dye and will be asked to lie still on the "scanning bed" for a period of 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* High risk ACS

  1. Angina [accelerating pattern or prolonged episode (> 20 minutes) or recurrent episode at rest or with minimal effort within preceding 24 hours]; and (13)
  2. Elevated Troponin - T (≥0.1 ug/L) or ECG changes consistent with ischemia [ST depression ≥ 0.1 mV, transient ST segment elevation ≥ 0.1 mV (< 20 minutes)]) (11;13)
* Planned conventional invasive coronary angiography

Exclusion Criteria:

* Age < 18 years or lack of consent
* Renal Insufficiency (GFR < 60 ml/min)
* Allergy to contrast agent
* Refractory angina requiring urgent/emergent coronary angiography (as per treating physician)
* Contraindication to radiation exposure (e.g. pregnancy)
* Uncontrolled HR
* Previous CABG or PCI/Stent
* Atrial fibrillation, frequent atrial or ventricular ectopy (> 1 / minute)
* Unable to perform 20 second breath-hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Operating Characteristics of CTA | 1 month

SECONDARY OUTCOMES:
To compare the accuracy of CTA to CICA in predicting the mode of revascularization (PCI versus CABG) in NSTE-ACS patients. | 1 month
To determine the number of "avoidable" CICA (i.e. those accurately designated to medical therapy or surgery with CTA). | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Carole Dennie, MD, Study Director — The Ottawa Hospital; Derek So, MD, Study Director — Ottawa Heart Institute Research Corporation; Chris Glvoer, MD, Study Director — Univeristy of Ottawa Heart Institute; Benjamin JW Chow, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- See also: University of Ottawa Heart Institute — http://www.ottawaheart.ca